CLINICAL TRIAL: NCT05777304
Title: Wearable Sensors and Machine Learning: a Technological Approach to Biomechanical Risk Assessment in Lifting Tasks
Brief Title: Wearable Sensors and Machine Learning for the Assessment of Biomechanical Risk in Lifting Tasks
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Edda Capodaglio, Principal Investigator, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2475
Record Dates: First submitted 2023-03-02; First posted 2023-03-21 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Wearable Devices
Keywords: inertial measurement units; Accelerometers; Ergonomics; Exposure assessment; Lifting; Work-related musculoskeletal disorders; Machine learning; Digital signal processing; Risk prediction
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: wearable device — IMU sensors and EMG sensors

SUMMARY:
Lifting loads can cause work-related musculoskeletal disorders. The National Institute for Occupational Safety and Health (NIOSH) established a methodology for assessing lifting actions by means of a quantitative method based on intensity, duration, frequency, and other geometrical characteristics of lifting. Body-worn inertial sensor technology provides a number of opportunities to advance the safety and health of workers engaged in physical work. Motion-tracking systems together with Machine learning (ML) algorithms are used in the ergonomic field for biomechanical risk assessment by means of data acquired by wearable inertial systems. The investigators posed the question whether it is possible to classify lifting tasks belonging to different risk classes according to the value of LI using a machine learning approach by means of features extracted from raw signals. Aim of this study was to develop and validate, through ML algorithms, a non-invasive detection system of kinetic-kinematic parameters using IMU and EMG sensors, for the ergonomic assessment of the risk associated with a load lifting activity.

DETAILED DESCRIPTION:
The study envisages the voluntary enrollment of healthy subjects, referring to treatment clinics for work-related pathologies (excluding subjects aged <18 or > 65 years, and those with musculoskeletal pathologies or other disabling pathologies in progress), to carry out two repeated lifting tests. The two tests are set up to correspond respectively to the two NIOSH risk classes (LI<1, NO RISK; and LI>1, RISK). The IMU sensors provide wirelessly a series of data from which it is intended to extract a number of features (feature extraction) that have a high predictive power, through the digital signal processing technique using dedicated software (i.e. Matlab, SPSS). In a second step, data obtained from EMG sensors will be added to the analysis. Among the different artificial intelligence algorithms, the investigator will look for those most able to discriminate the various risk classes on the basis of the parameters extracted from the signals detected during the motor task.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* subjects with musculoskeletal pathologies or other disabling pathologies in progress

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteer referring to treatment clinics for work-related pathologies
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Validation of the proposed strategy to assess the risk of lifting activities, according to RNLE | first year
  accuracy degree and AucRoc

CONTACTS AND LOCATIONS:
Overall Officials: Edda Capodaglio, PhD, Principal Investigator — ICS Maugeri IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Donisi L, Cesarelli G, Capodaglio E, Panigazzi M, D'Addio G, Cesarelli M, Amato F. A Logistic Regression Model for Biomechanical Risk Classification in Lifting Tasks. Diagnostics (Basel). 2022 Oct 29;12(11):2624. doi: 10.3390/diagnostics12112624. PMID 36359468
- [Result] Donisi L, Cesarelli G, Pisani N, Ponsiglione AM, Ricciardi C, Capodaglio E. Wearable Sensors and Artificial Intelligence for Physical Ergonomics: A Systematic Review of Literature. Diagnostics (Basel). 2022 Dec 5;12(12):3048. doi: 10.3390/diagnostics12123048. PMID 36553054
- [Result] Donisi L, Capodaglio EM, Amitrano F, Cesarelli G, Pagano G, D'Addio G. A multiple linear regression approach to extimate lifted load from features extracted from inertial data. G Ital Med Lav Ergon. 2021 Dec;43(4):373-378. PMID 35049162
- [Result] Donisi L, Cesarelli G, Coccia A, Panigazzi M, Capodaglio EM, D'Addio G. Work-Related Risk Assessment According to the Revised NIOSH Lifting Equation: A Preliminary Study Using a Wearable Inertial Sensor and Machine Learning. Sensors (Basel). 2021 Apr 7;21(8):2593. doi: 10.3390/s21082593. PMID 33917206